CLINICAL TRIAL: NCT01606683
Title: Impact of Infant Feeding on Newborn Metabolomic Profile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinz Italia SpA (Industry)
Collaborators: Fondazione IRCCS Policlinico San Matteo di Pavia (Other); University of Cagliari (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: PLA-LENI-09 - SUBSTUDY 1
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Formula Feeding of Healthy Full Term Infants; Breast Feeding of Healthy Full Term Infants
Keywords: Acidified milk; Beta-palmitate; Bifidobacteria; Breastfeeding; Infant formula; Galacto-oligosaccharides; Growth; Infants; Metabolomics; Prebiotics
MeSH Terms: conditions — Breast Feeding | interventions — Infant Formula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- GROUP 1 (Experimental): Infant formula supplemented with with functional ingredients (galacto-oligosaccharides, beta-palmitate, fermented milk). Infant formula with functional ingredients is in compliance with Directive 2006/141/CE on infant formulae and follow-on formulae.
  Interventions: Other: Infant formula with GOS, beta-palmitate, acidified milk
- GROUP 2 (Other): Standard infant formula, in compliance with Directive 2006/141/CE on infant formulae and follow-on formulae, without functional ingredients.
  Interventions: Other: Standard infant formula without functional ingredients
- CONTROL GROUP (Other): Breast milk
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Infant formula with GOS, beta-palmitate, acidified milk — Infant formula supplemented with functional ingredients (galacto-oligosaccharides, beta-palmitate, acidified milk.
  Infant formula with functional ingredients is in compliance with Directive 2006/141/CE on infant formulae and follow-on formulae.
  Arms: GROUP 1
Other: Standard infant formula without functional ingredients — Standard infant formula, in compliance with Directive 2006/141/CE on infant formulae and follow-on formulae, without functional ingredients.
  Arms: GROUP 2
Other: No intervention
  Arms: CONTROL GROUP

SUMMARY:
The purpose of this study is the evaluation with untargeted modalities, of the urine metabolomic profile in a group of infants fed with a standard formula, a group of infants fed with a formula supplemented with functional ingredients and a group of breast-fed infants.

DETAILED DESCRIPTION:
Metabolomics is of particular interest in the field of nutrition, since nutrients interact with a number of targets, metabolic pathways and functions.

A suitable biofluid to study nutrient intake is urine, which is the most commonly used biological sample for metabolomic analysis and can be collected with simple and non-invasive methods.

Up to now, no studies have investigated healthy term infants metabolome and its modulation according to different dietary regimens such as formula-feeding or breastfeeding.

The aim of this study is to evaluate, with untargeted modalities, the urine metabolomic profile of a group of infants fed with a standard formula, a group of infants fed with a formula supplemented with functional ingredients and a group of breast-fed infants.

Formula-fed infants participate to PLA-LENI-09 study (NCT01197365). We have included also a control group of breast-fed infants, as, from a scientific point of view, they represent the "gold standard" and no data are available on their metabolomic profile.

ELIGIBILITY:
Inclusion Criteria:

* Infants being exclusively either breastfed or formula-fed by the 21st day of life
* Infants of both sexes born with natural or caesarian delivery
* Gestational age between 37 and 42 completed weeks
* Birth weight between 10th and 90th percentile of birth weight for gestational age, according to the North-Italian growth charts
* Single birth
* Caucasian parents

Exclusion Criteria:

* Infants with genetic and/or congenital diseases
* Infants receiving antibiotic therapy
* Infants with neonatal diseases requiring hospitalisation for longer than 7 days
* Infants at risk for atopy and/or having familial history for atopy
* Mothers with metabolic or chronic diseases
* Infant selected for another clinical study
* Parents refusing to sign a written informed consent

Max Age: 21 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2012-04; Primary Completion 2013-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Metabolite patterns associated with different dietary regimens | At enrolment, after 60 and 135 days of life
  Urine will be analysed using 1H-NMR. Data will be analyzed through the use of software products to enable the discovery of hundreds of different metabolites involved in multiple pathways and connected with different conditions. The metabolites on which the univariate analysis will be performed are the most important revealed by the multivariate analysis (VIP variables) and Student's statistical test will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Stronati, Prof., Principal Investigator — FONDAZIONE IRCCS POLICLINICO "SAN MATTEO" - STRUTTURA COMPLESSA DI NEONATOLOGIA, PATOLOGIA NEONATALE E TERAPIA INTENSIVA
Locations (1):
- Fondazione Irccs Policlinico "San Matteo" - Struttura Complessa Di Neonatologia, Patologia Neonatale E Terapia Intensiva, Pavia, PV, Italy

REFERENCES:
- [Background] Goodacre R, Vaidyanathan S, Dunn WB, Harrigan GG, Kell DB. Metabolomics by numbers: acquiring and understanding global metabolite data. Trends Biotechnol. 2004 May;22(5):245-52. doi: 10.1016/j.tibtech.2004.03.007. No abstract available. PMID 15109811
- [Background] Ryan D, Robards K. Metabolomics: The greatest omics of them all? Anal Chem. 2006 Dec 1;78(23):7954-8. doi: 10.1021/ac0614341. No abstract available. PMID 17134127
- [Background] Fanos V, Barberini L, Antonucci R, Atzori L. Metabolomics in neonatology and pediatrics. Clin Biochem. 2011 May;44(7):452-454. doi: 10.1016/j.clinbiochem.2011.03.006. No abstract available. PMID 22036322
- [Background] Atzori L, Antonucci R, Barberini L, Griffin JL, Fanos V. Metabolomics: a new tool for the neonatologist. J Matern Fetal Neonatal Med. 2009;22 Suppl 3:50-3. doi: 10.1080/14767050903181500. PMID 19701858
- [Background] Goodacre R. Metabolomics of a superorganism. J Nutr. 2007 Jan;137(1 Suppl):259S-266S. doi: 10.1093/jn/137.1.259S. PMID 17182837
- [Background] Nicholson JK, Wilson ID. Opinion: understanding 'global' systems biology: metabonomics and the continuum of metabolism. Nat Rev Drug Discov. 2003 Aug;2(8):668-76. doi: 10.1038/nrd1157. No abstract available. PMID 12904817
- [Background] Nicholson JK, Holmes E, Lindon JC, Wilson ID. The challenges of modeling mammalian biocomplexity. Nat Biotechnol. 2004 Oct;22(10):1268-74. doi: 10.1038/nbt1015. PMID 15470467
- [Background] Carraro S, Giordano G, Reniero F, Perilongo G, Baraldi E. Metabolomics: a new frontier for research in pediatrics. J Pediatr. 2009 May;154(5):638-44. doi: 10.1016/j.jpeds.2009.01.014. No abstract available. PMID 19364557
- [Background] Janeckova H, Hron K, Wojtowicz P, Hlidkova E, Baresova A, Friedecky D, Zidkova L, Hornik P, Behulova D, Prochazkova D, Vinohradska H, Peskova K, Bruheim P, Smolka V, Stastna S, Adam T. Targeted metabolomic analysis of plasma samples for the diagnosis of inherited metabolic disorders. J Chromatogr A. 2012 Feb 24;1226:11-7. doi: 10.1016/j.chroma.2011.09.074. Epub 2011 Oct 4. PMID 22018716
- [Background] Atzori L, Antonucci R, Barberini L, Locci E, Cesare Marincola F, Scano P, Cortesi P, Agostiniani R, Weljie A, Lai A, Fanos V. 1H NMR-based metabolic profiling of urine from children with nephrouropathies. Front Biosci (Elite Ed). 2010 Jan 1;2(2):725-32. doi: 10.2741/e132. PMID 20036916
- [Background] Atzori L, Antonucci R, Barberini L, Locci E, Marincola FC, Scano P, Cortesi P, Agostiniani R, Defraia R, Weljie A, Gazzolo D, Lai A, Fanos V. 1H NMR-based metabolomic analysis of urine from preterm and term neonates. Front Biosci (Elite Ed). 2011 Jun 1;3(3):1005-12. doi: 10.2741/e306. PMID 21622109
- [Background] Ciccarelli S, Atzori L, Noto A, Barberini L, Fanos V, Caramia G, Agostino R. Spontaneous vs cesarean delivery: a metabolomic point of view. J Matern Fetal Neonatal Med 24(S(2):1-2, 2011.
- [Background] Scalbert A, Brennan L, Fiehn O, Hankemeier T, Kristal BS, van Ommen B, Pujos-Guillot E, Verheij E, Wishart D, Wopereis S. Mass-spectrometry-based metabolomics: limitations and recommendations for future progress with particular focus on nutrition research. Metabolomics. 2009 Dec;5(4):435-458. doi: 10.1007/s11306-009-0168-0. Epub 2009 Jun 12. PMID 20046865
- [Background] Gibney MJ, Walsh M, Brennan L, Roche HM, German B, van Ommen B. Metabolomics in human nutrition: opportunities and challenges. Am J Clin Nutr. 2005 Sep;82(3):497-503. doi: 10.1093/ajcn.82.3.497. PMID 16155259
- [Background] Walsh MC, Brennan L, Malthouse JP, Roche HM, Gibney MJ. Effect of acute dietary standardization on the urinary, plasma, and salivary metabolomic profiles of healthy humans. Am J Clin Nutr. 2006 Sep;84(3):531-9. doi: 10.1093/ajcn/84.3.531. PMID 16960166
- [Background] Phipps AN, Stewart J, Wright B, Wilson ID. Effect of diet on the urinary excretion of hippuric acid and other dietary-derived aromatics in rat. A complex interaction between diet, gut microflora and substrate specificity. Xenobiotica. 1998 May;28(5):527-37. doi: 10.1080/004982598239443. PMID 9622854
- [Background] Bell JD, Sadler PJ, Morris VC, Levander OA. Effect of aging and diet on proton NMR spectra of rat urine. Magn Reson Med. 1991 Feb;17(2):414-22. doi: 10.1002/mrm.1910170213. PMID 1829498
- [Background] Zhang X, Yap Y, Wei D, Chen G, Chen F. Novel omics technologies in nutrition research. Biotechnol Adv. 2008 Mar-Apr;26(2):169-76. doi: 10.1016/j.biotechadv.2007.11.002. Epub 2007 Nov 19. PMID 18164161
- [Background] Bertram HC, Hoppe C, Petersen BO, Duus JO, Molgaard C, Michaelsen KF. An NMR-based metabonomic investigation on effects of milk and meat protein diets given to 8-year-old boys. Br J Nutr. 2007 Apr;97(4):758-63. doi: 10.1017/S0007114507450322. PMID 17349089